CLINICAL TRIAL: NCT01077986
Title: A Phase I/ II, Non-randomized, Feasibility/ Safety and Efficacy Study of the Combination of Everolimus, Cetuximab and Capecitabine in Patients With Metastatic Pancreatic Cancer
Brief Title: Everolimus, Cetuximab and Capecitabine in Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.W. Wilmink, Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCmedonc08/345
Record Dates: First submitted 2010-02-25; First posted 2010-03-02 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: mTOR inhibition; EGFR inhibition; pancreatic cancer; pharmacodynamics
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Cetuximab; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Capecitabine — Capecitabine will be administered for 14 days in a 3 weekly cycle, starting on day 8.
  Other Names: Xeloda
Drug: Cetuximab — Cetuximab will be administered weekly, starting at day 8.
  Other Names: Erbitux
Drug: Everolimus — Everolimus will be administered daily, starting on day 1.
  Other Names: certican

SUMMARY:
In this study the investigators want to determine the activity and safety of concurrent interruption of the MAPK and PI3K pathways by EGFR and mTOR inhibition in patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This phase I/II non randomized single center study will be performed as a two step design. Part I is dose finding, whereby dose escalations will be performed for everolimus and capecitabine. Part II is the efficacy study. At the MTD doses in part II biomarker studies will be performed in blood and tumor tissue. Study design phase I part: The first week patients will be treated with everolimus alone. Capecitabine will be administered for 14 days in a 3 weekly cycle, starting on day 8. Cetuximab will be administered weekly, starting at day 8. The dose is fixed for cetuximab during study treatment, whereas the doses of everolimus and capecitabine will differ per dose level. First dose level: Everolimus 5 mg daily continuously, Capecitabine 600 mg/m2 bid for 2 weeks every 3 weeks, Cetuximab 400mg/m2 (120 min infusion) first dose, thereafter 250 mg/m2 (60 min infusion) weekly. Second dose level: Everolimus 10 mg daily continuously, Capecitabine 600 mg/m2 bid for 2 weeks every 3 weeks, Cetuximab 400mg/m2 (120 min infusion) first dose, thereafter 250 mg/m2 (60 min infusion) weekly. Third dose level: Everolimus 10 mg daily continuously, Capecitabine 800 mg/m2 bid for 2 weeks every 3 weeks, Cetuximab 400mg/m2 (120 min infusion) first dose, thereafter 250 mg/m2 (60 min infusion) weekly. Study design phase II part At the MTD 14-25 patients with pancreatic cancer will be included. In the phase II part, everolimus will be administered during one week before start of cetuximab. At day 8 the first dose of cetuximab will be administered. Capecitabine will be started one week thereafter. This enables us to perform pharmacodynamic studies to assess biomarker changes during the different phases of treatment. Everolimus will be administered continuously in a dose of 5 or 10 mg orally once daily (dependent on MTD from part 1). Capecitabine will be administered orally in a dose of 400 - 800 mg/m2 twice daily for 14 days followed by one week rest (dependent on MTD from part 1). Patients will receive cetuximab infusions via an infusion pump, with an initial dose of 400 mg/m² (over 120 min) and subsequent weekly infusions of 250 mg/m² (over 60 min), starting day 8.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed content obtained prior to treatment
* Cytological or histological confirmed adenocarcinoma of the pancreas
* Metastatic pancreatic cancer
* Measurable lesion according to RECIST criteria
* ECOG/ WHO performance 0-2
* Age > 18 years
* Life expectancy > 3 months
* Adequate renal function (creatinine < 150 µmol/L)
* Adequate liver function (bilirubin < 1.5 times upper limit of normal, ALAT or ASAT < 5.0 times upper limit of normal in case of liver metastases and < 2.5 the upper limit of normal in absence of liver metastases
* Adequate bone marrow function (WBC > 3.0 x 10 9/L, platelets > 100 x 10 9/L)
* Mentally, physically, and geographically able to undergo treatment and follow up

Exclusion Criteria:

* Clinical or radiological evidence of CNS metastases
* Pregnancy (positive serum pregnancy test) and lactation
* Serious concomitant systemic disorder that would compromise the safety of the patient, at the discretion of the investigator
* Patients who have any severe and/or uncontrolled medical conditions
* Previous treatment with an mTOR inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
phase I part: assessment of the dose limiting toxicity | During treatment: assessments on day 1 every cycle (3 weeks). After treatment: every 3 months during the first 2 years, and every 6 months thereafter
phase II part: response rate | Assessments after every 3 cycles (9 weeks).

SECONDARY OUTCOMES:
Time to treatment failure | Every 3 months during the first 2 years, and every 6 months thereafter.
Overall survival | Every 3 months during the first 2 years, and every 6 months thereafter.
Toxicity profile | During treatment: assessments on day 1 every cycle (3 weeks). After treatment: every 3 months during the first 2 years, and every 6 months thereafter.
Pharmacodynamics: biomarkers in blood and tumor tissue | Day 1, 8 and 22 during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke Wilmink, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands